CLINICAL TRIAL: NCT00957541
Title: Clinical Evaluation of the Physiological Diagnosis Function in the Paradym CRT Device
Brief Title: Evaluation of a Diagnostic Feature in a Cardiac Resynchronization Therapy (CRT) Device
Acronym: CLEPSYDRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ELA Medical, Inc. (Industry)
Collaborators: LivaNova (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: ITSY02
Record Dates: First submitted 2009-08-10; First posted 2009-08-12 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-05

CONDITIONS: Congestive Heart Failure
Keywords: NYHA Class III or IV; Implantable Cardiac Defibrillator; Cardiac Resynchronization Therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CRT Therapy (Experimental): All patients will receive CRT therapy with the Physiological Diagnosis (PhD) feature enabled.
  Interventions: Device: Paradym CRT + Physiological Diagnosis (PhD)

INTERVENTIONS:
Device: Paradym CRT + Physiological Diagnosis (PhD) — All subjects will undergo CRT therapy with the Physiological Diagnosis (PhD) feature enabled.

SUMMARY:
The purpose of this study is to evaluate the performance of a new sensor-based diagnostic feature, which has been implemented in a cardiac resynchronization therapy (CRT) device. This trial will study the effectiveness of the diagnostic feature to detect heart failure events in medically stable, ICD-indicated, congestive heart failure patients.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the performance of a new sensor-based diagnostic feature, which has been implemented in a cardiac resynchronization therapy (CRT) device. This trial will study the effectiveness of the diagnostic feature to detect heart failure events in medically stable, ICD-indicated, congestive heart failure patients. The ability of the diagnostic feature to 'detect' and 'predict' heart failure events will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Subject eligible for implantation of a CRT-D device according to current available guidelines for cardiac resynchronization therapy
* Subject has severe heart failure (NYHA Class III or IV)
* Subject has experienced at least one heart failure event within six months prior to enrollment
* Subject continues to have heart failure symptoms despite receiving optimal medical therapy
* Schedule for implant of a PARADYM CRT-D (Model 8770)
* Subject has signed and dated an informed consent form

Exclusion Criteria:

* Any contraindication for standard cardiac pacing
* Any contraindication for ICD therapy
* Abdominal implantation site
* Hypertrophic or obstructive cardiomyopathy
* Acute myocarditis
* Unstable coronary symptoms (unstable angina or myocardial infarction) within the last month
* Recent (within the last month) or planned cardiac revascularization or coronary angioplasty
* Correctable valvular disease that is the primary cause of heart failure
* Mechanical tricuspid valve
* Receiving continuous intra-venous infusion of positive inotropic therapy or intermittent therapy (intravenous infusion) more than twice per week
* Heart transplant recipient
* Renal insufficiency requiring dialysis
* Already included in another clinical study
* Life expectancy less than 12 months
* Inability to understand the purpose of the study or refusal to cooperate
* Inability or refusal to provide informed consent or HIPAA
* Unavailability for scheduled follow-up at the implanting center
* Known sensitivity to 1mg dexamethasone sodium phosphate (DSP)
* Under guardianship
* Age of less than 18 years
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2009-09; Primary Completion 2011-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Sensitivity of diagnostic feature in detecting heart failure events (using the device) in comparison to clinical heart failure events experienced by the patient (as classified by an independent committee). | Thirteen months
Mean number of false positives per patient per year. | Thirteen Months

CONTACTS AND LOCATIONS:
Locations (1):
- Mountain Vista Hospital, Mesa, Arizona, United States

REFERENCES:
- [Background] Auricchio A, Brugada J, Ellenbogen KA, Gold MR, Leyva F; CLEPSYDRA investigators. Assessment of a novel device-based diagnostic algorithm to monitor patient status in moderate-to-severe heart failure: rationale and design of the CLEPSYDRA study. Eur J Heart Fail. 2010 Dec;12(12):1363-71. doi: 10.1093/eurjhf/hfq170. Epub 2010 Oct 14. PMID 20947571